CLINICAL TRIAL: NCT03009344
Title: A Phase 1 Study of Tazemetostat in Patients With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: A Study of Tazemetostat in Participants With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7438-J081-106
Record Dates: First submitted 2016-12-30; First posted 2017-01-04 (Estimated); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-04

CONDITIONS: Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Keywords: relapsed or refractory B-cell non-Hodgkin's lymphoma; tazemetostat; Japan; E7438
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tazemetostat 800 mg (Experimental): Participants will receive oral tazemetostat at a starting dose of 800 milligrams (mg) as a single dose (Cycle 0) and 800 mg twice a day as continuous dosing (Cycle 1 and later) (Cycle 0 duration=4 days) (Cycle 1 and later duration= 28 days).
  Interventions: Drug: Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat tablets.

SUMMARY:
This is a multicenter, single-arm, open-label, Phase 1 study to assess the tolerability, safety, pharmacokinetics, and preliminary anti-tumor activity of tazemetostat in participants with relapsed or refractory B-cell non-Hodgkin's lymphoma (NHL).

ELIGIBILITY:
Inclusion Criteria:

* Participants with histological diagnosis of B-cell non-Hodgkin's lymphoma
* Participant who has measurable disease
* Participant who had previous therapy with systemic chemotherapy and/or antibody therapy
* Participant who had progressive disease (PD) or did not have a response (complete response [CR] or partial response [PR]) in previous systemic therapy, or relapsed or progressed after previous systemic therapy
* Participant with Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Participant with life expectancy of ≥3 months from starting study drug administration
* Participant with adequate renal, bone marrow, and liver function
* Participant with left ventricular ejection fraction (LVEF) > 50%
* Male and female participant ≥20 years of age at the time of informed consent
* Participant who has provided written consent to participate in the study

Exclusion Criteria:

* Participant with prior exposure to EZH2 inhibitor
* Participant with a history or a presence of central nerves invasion
* Participant with allogeneic stem cell transplantation
* Participant with medical need for the continued use of potent or moderate inhibitors of CYP3A or P-gp, or potent or moderate inducer of CYP3A (including St. John's wort).
* Participant with significant cardiovascular impairment
* Participant with prolongation of corrected QT interval using Fridericia's formula (QTcF) to > 480 milliseconds (msec)
* Participant with venous thrombosis or pulmonary embolism within the last 3 months before starting study drug
* Participant with complications of hepatic cirrhosis, interstitial pneumonia, or pulmonary fibrosis
* Participant with active infection requiring systemic therapy
* Women of childbearing potential or man of impregnate potential who don't agree to use a medically effective method for contraception for periods from before informed consent to during the clinical study and 30 days later from last administration of study drug
* Woman who are pregnant or breastfeeding
* Participant who were deemed as inappropriate to participate in the study by the investigator or sub-investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Eisai Trial Site, Isehara, Kanagawa
  - Eisai Trial Site, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Japan from 10 January 2017 to 17 June 2020.
Pre-assignment Details: A total of 7 participants were screened and enrolled to receive study treatment.
Groups:
- Tazemetostat 800 mg: Participants received tazemetostat 800 milligram (mg) tablets, orally on Day 1 of Cycle 0 and 800 mg tablets, orally, twice daily as continuous dosing in Cycle 1 and later cycles until disease progression (PD), development of unacceptable toxicity, participant request to discontinue, withdrawal of consent, or study termination by the sponsor (up to 39 months). Cycle 0 duration was 4 days, Cycle 1 and later cycles duration was 28 days.
Period: Overall Study
Arm/Group | Tazemetostat 800 mg
Started | 7
Completed | 0
Not Completed | 7
Not completed — Lack of Efficacy | 5
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The safety/efficacy analysis set included all participants who received at least 1 administration of the study drug.
Groups:
- Tazemetostat 800 mg: Participants received tazemetostat 800 mg tablets, orally on Day 1 of Cycle 0 and 800 mg tablets, orally, twice daily as continuous dosing in Cycle 1 and later cycles until PD, development of unacceptable toxicity, participant request to discontinue, withdrawal of consent, or study termination by the sponsor (up to 39 months). Cycle 0 duration was 4 days, Cycle 1 and later cycles duration was 28 days.
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs as per National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03) were defined as: 1) Grade 4 neutropenia for greater than (>) 7 days; 2) greater than or equal to (>=) Grade 3 febrile neutropenia; 3) Grade 4 thrombocytopenia and Grade 3 thrombocytopenia with bleeding; 4) Grade 4 anemia or anemia requiring erythrocyte transfusion; 5) >=Grade 3 nausea, vomiting, or diarrhea that persisted >7 days despite maximal medical therapy; 6) >=Grade 3 non-hematological laboratory abnormalities with clinical symptoms that persisted >7 days; 7) Other Grade 3 toxicity lasting >7 days or Grade 4 non-hematological toxicity of any duration; 8) Failure to administer >=75 percent (%) of the planned administration number of study drug in Cycle 1 as a result of treatment-related toxicity. Here, number of participants who had DLT were reported.
Time Frame: Cycle 0 and Cycle 1 (Cycle 0=4 days, Cycle 1=28 days)
Population: DLT analysis set included all participants who completed treatment Cycles 0 and 1 without major protocol deviations with at least 75% of treatment compliance in Cycle 1 and were assessed for DLT, and participants who experienced DLT during Cycles 0 and 1. Participants with less than 75% treatment compliance in Cycle 1 due to a reason other than toxicity up to Cycle 1 Day 28 were not included in this analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAE was defined as an adverse event (AE) that emerged during time from first dose to 30 days following last dose of drug, having been absent at pretreatment or reemerged during treatment, having been present at pretreatment but stopped before treatment, or worsened in severity during treatment relative to pretreatment state, when AE was continuous. Number of participants with TEAEs were reported based on their safety assessments of laboratory tests, physical examination, regular measurement of vital signs, body weight, echocardiograms/multigated acquisition (MUGA) scans to assess left ventricular ejection fraction, eastern cooperative oncology group-performance status (ECOG-PS) and electrocardiograms parameter values. SAE was defined as untoward medical occurrence that at any dose resulted in death; was life threatening; resulted in persistent or significant disability; was congenital anomaly or medically important due to other reasons than above mentioned criteria.
Time Frame: From the date of first dose up to 30 days after the last dose of study drug (up to 40 months)
Population: The safety analysis set included all participants who received at least 1 administration of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
Participants
  TEAEs | 7
  SAEs | 2

3. Secondary Outcome: Cmax: Maximum Plasma Concentration of Tazemetostat and Its Metabolite ER-897387
Time Frame: Cycle 0 Day 1: 0-72 hours post-dose (Cycle 0 length=4 days)
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 administration of the study drug and had sufficient PK data to derive at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
nanogram per milliliter (ng/mL)
  Tazemetostat | 988 (62.1)
  ER-897387 | 790 (78.8)

4. Secondary Outcome: Tmax: Time to Reach Maximum Plasma Concentration (Cmax) of Tazemetostat and Its Metabolite ER-897387
Time Frame: Cycle 0 Day 1: 0-72 hours post-dose (Cycle 0 length=4 days)
Population: The PK analysis set included all participants who received at least 1 administration of the study drug and had sufficient PK data to derive at least 1 PK parameter.
Measure: Median (Full Range); unit: hours
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
hours
  Tazemetostat | 1.97 [0.95 to 4.08]
  ER-897387 | 1.97 [1.12 to 4.08]

5. Secondary Outcome: AUC(0-12 Hours): Area Under the Plasma Concentration-time Curve From Time Zero to 12 Hours Post-dose of Tazemetostat and Its Metabolite ER-897387
Time Frame: Cycle 0 Day 1: 0-12 hours post-dose (Cycle 0 length=4 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
nanogram*hour per milliliter (ng*h/mL)
  Tazemetostat | 4080 (61.3)
  ER-897387 | 4500 (72.4)

6. Secondary Outcome: AUC(0-t Hours): Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration of Tazemetostat and Its Metabolite ER-897387
Time Frame: Cycle 0 Day 1: 0-72 hours post-dose (Cycle 0 length=4 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
ng*h/mL
  Tazemetostat | 5180 (63.6)
  ER-897387 | 6540 (75.3)

7. Secondary Outcome: AUC(0-infinity): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity of Tazemetostat and Its Metabolite ER-897387
Time Frame: Cycle 0 Day 1: 0-72 hours post-dose (Cycle 0 length=4 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
ng*h/mL
  Tazemetostat | 5220 (63.2)
  ER-897387 | 6570 (74.9)

8. Secondary Outcome: Lambda z: Terminal Phase Elimination Rate Constant of Tazemetostat and Its Metabolite ER-897387
Description: Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: Cycle 0 Day 1: 0-72 hours post-dose (Cycle 0 length=4 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
per hour
  Tazemetostat | 0.0925 (17.9)
  ER-897387 | 0.0794 (16.9)

9. Secondary Outcome: T1/2: Terminal Half-life of Tazemetostat and Its Metabolite ER-897387
Time Frame: Cycle 0 Day 1: 0-72 hours post-dose (Cycle 0 length=4 days); Cycle 1 Day 15: 0-12 hours post-dose (Cycle 1 length=28 days)
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
hour
  Tazemetostat (Cycle 0 Day 1) | 7.76 [5.24 to 9.32]
  Tazemetostat (Cycle 1 Day 15) | 4.10 [2.40 to 8.31]
  ER-897387 (Cycle 0 Day 1) | 8.68 [6.52 to 10.7]
  ER-897387 (Cycle 1 Day 15) | 3.55 [3.22 to 9.58]

10. Secondary Outcome: CL/F: Apparent Total Body Clearance of Tazemetostat
Time Frame: Cycle 0 Day 1: 0-72 hours post-dose (Cycle 0 length=4 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
liter per hour (L/h) | 153 (63.2)

11. Secondary Outcome: Vz/F: Apparent Volume of Distribution at Terminal Phase of Tazemetostat
Description: Vz/F for Cycle 0 Day 1 was calculated as Dose divided by ([lambda z]*[AUC0-infinity]) and for Cycle 1 Day 15 was calculated as Dose divided by ([lambda z]*[AUC0-tau]).
Time Frame: as for outcome 9
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
liter (L)
  Cycle 0 Day 1 | 1660 (64.1)
  Cycle 1 Day 15 | 1170 (93.0)

12. Secondary Outcome: MRT: Mean Residence Time of Tazemetostat and Its Metabolite ER-897387
Description: MRT of tazemetostat and its metabolite ER-897387 was calculated as MRT=AUMC(0-infinity)/AUC(0-infinity), where AUMC(0-infinity) was the area under the first moment curve extrapolated to infinity and AUC(0-infinity) was area under the concentration-time curve from zero time extrapolated to infinite time.
Time Frame: Cycle 0 Day 1: 0-72 hours post-dose (Cycle 0 length=4 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
hours
  Tazemetostat | 8.25 (29.3)
  ER-897387 | 10.7 (31.0)

13. Secondary Outcome: AUC(0-tau): Area Under the Plasma Concentration-time Curve Over the Dosing Interval of Tazemetostat and Its Metabolite ER-897387
Time Frame: Cycle 1 Day 15: 0-12 hours post-dose (Cycle 1 length=28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
ng*h/mL
  Tazemetostat | 4220 (42.6)
  ER-897387 | 10200 (39.1)

14. Secondary Outcome: Css,Av: Average Steady State Plasma Concentration of Tazemetostat and Its Metabolite ER-897387
Time Frame: Cycle 1 Day 15: 0-12 hours post-dose (Cycle 1 length=28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
ng/mL
  Tazemetostat | 351 (42.7)
  ER-897387 | 852 (39.0)

15. Secondary Outcome: Css,Max: Maximum Steady State Plasma Concentration of Tazemetostat and Its Metabolite ER-897387
Time Frame: Cycle 1 Day 15: 0-12 hours post-dose (Cycle 1 length=28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
ng/mL
  Tazemetostat | 1170 (51.6)
  ER-897387 | 1800 (47.4)

16. Secondary Outcome: Css,Min: Minimum Steady State Plasma Concentration of Tazemetostat and Its Metabolite ER-897387
Time Frame: Cycle 1 Day 15: 0-12 hours post-dose (Cycle 1 length=28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
ng/mL
  Tazemetostat | 88.4 (43.8)
  ER-897387 | 293 (46.7)

17. Secondary Outcome: PTF: Peak-trough Fluctuation Ratio of Tazemetostat and Its Metabolite ER-897387
Description: The PTF within complete dosing interval at steady state, calculated as PTF (%) = ([Cmax - Cmin]/Cav) multiplied by 100. Here, Cmin means the minimum plasma concentration, Cmax means the maximum plasma concentration and Cav means the average plasma concentration of drug and metabolite.
Time Frame: Cycle 1 Day 15: 0-12 hours post-dose (Cycle 1 length=28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage fluctuation
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
percentage fluctuation
  Tazemetostat | 303 (40.8)
  ER-897387 | 171 (39.8)

18. Secondary Outcome: Tss,Max: Time to Reach the Maximum Plasma Concentration (Cmax) at Steady State of Tazemetostat and Its Metabolite ER-897387
Time Frame: Cycle 1 Day 15: 0-12 hours post-dose (Cycle 1 length=28 days)
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
hours
  Tazemetostat | 1.05 [0.88 to 2.03]
  ER-897387 | 1.07 [0.88 to 2.03]

19. Secondary Outcome: CLss/F: Apparent Total Body Clearance of Tazemetostat at Steady State
Time Frame: Cycle 1 Day 15: 0-12 hours post-dose (Cycle 1 length=28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
L/h | 190 (42.6)

20. Secondary Outcome: Rac (Cmax): Accumulation Ratio of Cmax for Tazemetostat and Its Metabolite ER-897387
Description: Rac (Cmax) was calculated as the ratio of maximum observed concentration at steady state (Css,max) on Cycle 1 Day 15 divided by Cmax on Cycle 0 Day 1.
Time Frame: Cycle 0 Day 1: 0-72 hours post-dose (Cycle 0 length=4 days) and Cycle 1 Day 15: 0-12 hours post-dose (Cycle 1 length=28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
ratio
  Tazemetostat | 1.19 (56.7)
  ER-897387 | 2.28 (59.9)

21. Secondary Outcome: Rac (AUC): Accumulation Ratio of AUC for Tazemetostat and Its Metabolite ER-897387
Description: Rac (AUC) was calculated as the ratio of AUC(0-tau) on Cycle 1 Day 15 divided by AUC(0-12 hours) on Cycle 0 Day 1.
Time Frame: as for outcome 20
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
ratio
  Tazemetostat | 1.04 (37.6)
  ER-897387 | 2.27 (58.5)

22. Secondary Outcome: Rss: Steady State Accumulation Ratio of Tazemetostat and Its Metabolite ER-897387
Description: Rss was calculated as the ratio of AUC(0-tau) on Cycle 1 Day 15 divided by AUC(0-infinity) on Cycle 0 Day 1.
Time Frame: as for outcome 20
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
ratio
  Tazemetostat | 0.809 (35.0)
  ER-897387 | 1.56 (53.1)

23. Secondary Outcome: Ae: Amount of Unchanged Drug Tazemetostat Excreted in Urine
Time Frame: as for outcome 9
Population: The PK analysis set included all participants who received at least 1 administration of the study drug and had sufficient PK data to derive at least 1 PK parameter. Here number analyzed "n" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
mg
  Cycle 0 Day 1: number analyzed (Participants) | 6
  Cycle 0 Day 1 | 15.1 (51.6)
  Cycle 1 Day 15 | 6.81 (33.7)

24. Secondary Outcome: Fe: Fraction of Tazemetostat Dose Excreted in Urine
Description: The fraction of dose excreted in urine was calculated as: Cumulative amount of unchanged drug excreted in urine (Ae)/Dose*100.
Time Frame: as for outcome 9
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
percentage of dose
  Cycle 0 Day 1: number analyzed (Participants) | 6
  Cycle 0 Day 1 | 1.89 (51.4)
  Cycle 1 Day 15 | 0.852 (33.8)

25. Secondary Outcome: CLR: Renal Clearance of Tazemetostat
Time Frame: as for outcome 9
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
L/h
  Cycle 0 Day 1: number analyzed (Participants) | 6
  Cycle 0 Day 1 | 2.62 (15.2)
  Cycle 1 Day 15 | 1.62 (25.6)

26. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response was assessed by investigator based on the Lugano Classification (CT-Based) response criteria. Objective response rate was defined as the percentage of participants who had a Best Overall Response (BOR) of complete response (CR) or partial response (PR). CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurred first (up to 39 months)
Population: The efficacy analysis set included all participants who received at least 1 administration of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tazemetostat 800 mg
Number analyzed (Participants) | 7
percentage of participants | 57.1 [18.4 to 90.1]

ADVERSE EVENTS:
Time Frame: From the date of first dose up to 30 days after the last dose of study drug (up to 40 months)
Description: The safety analysis set included all participants who received at least 1 administration of the study drug.
Arm/Group | Tazemetostat 800 mg
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tazemetostat 800 mg (N=7)
Intestinal perforation (Gastrointestinal disorders) | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tazemetostat 800 mg (N=7)
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
Dry eye (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Asthenia (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 5
Influenza (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Weight decreased (Investigations) | 1
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysgeusia (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Middle insomnia (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin swelling (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT03009344/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT03009344/SAP_001.pdf